CLINICAL TRIAL: NCT02133898
Title: The Use Of A Genetic Marker To Predict Response To L-Methylfolate As A Treatment For Depression
Brief Title: The Use Of L-Methylfolate As A Treatment For Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Pamlab, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB201400170
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Depression
Keywords: Depression; MTHFR; L-methylfolate
MeSH Terms: conditions — Depression | interventions — 5-methyltetrahydrofolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- L-methyfolate (Other): Single-arm open label administration of L-methylfolate 15mg once daily for 90 days
  Interventions: Other: L-methylfolate

INTERVENTIONS:
Other: L-methylfolate — L-methylfolate, an FDA approved medical food will be administered in 15 mg capsule form once daily for 90 days
  Other Names: Deplin

SUMMARY:
This is an open-label study assessing the efficacy of l-methylfolate as monotherapy in patients with mild to moderate major depressive disorder (MDD). The plan is to enroll 75 patients with mild to moderate MDD based on the Structured Clinical Interview for DSM-IV (SCID) that have a Hamilton Depression Rating Scale-24 (HDRS-24) score between 8-24. The investigators will collect genotype data on methylenetetrahydrofolate Reductase (MTHFR), MTR and MTRR in this patient population. Subjects will be able to receive their genotype results, on request, upon completion of the study. The investigators hypothesize that depressed patients will be more likely to have a mutation in the MTHFR gene

DETAILED DESCRIPTION:
Participation in the study will consist of the following visits and test:

Screening Visit will include being interviewed by a staff member to determine qualification. This interview will involve a thorough diagnostic interview that asks about different psychological feelings and It will also involve several rating scales that ask about depression, anxiety, obsessive compulsive disorder (OCD), and suicidality. The following scales will be conducted at this visit:

Structured Clinical Interview for Diagnostic and Statistical Manual for Mental Disorders-IV (DSM) (SCID-I) is a clinician-administered, semi-structured diagnostic interview for mental health disorders.

Hamilton Depression Rating Scale-24 (HAM-D) is a clinician-administered questionnaire designed to assess the severity of depression in adults.

Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered questionnaire which assesses the severity of symptoms of anxiety.

Yale-Brown Obsessive Compulsive Scale (YBOCS) is a clinician administered questionnaire to assess the severity of symptoms of obsessive compulsive disorder.

The Montreal Cognitive Assessment (MoCA) is a clinician administered cognitive screening tool to aid in the detection of mild cognitive impairment.

The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician-administered rating scale that quantifies the presence and severity of suicidal ideation and behavior.

Clinical Global Impression-Severity (CGI-S) is a 7-point clinician rating of severity of psychopathology.

Next, a physician will conduct a brief medical physical exam which includes: measuring blood pressure, pulse, and body weight, a current and past medical history and blood will be drawn. If you are a female of childbearing potential, a urine pregnancy test will be performed.

Baseline Visit The results of the laboratory tests performed at the screening visit will be reviewed. If eligibility is met, vital signs (blood pressure, heart rate, and weight) will be measured. Then a member of the research team will ask questions about current symptoms. The following scales will be conducted at this visit and at all remaining visits in the study: HAM-D, HAM-A, YBOCS, MoCA, C-SSRS, and the CGI-S.

Clinical Global Impression-Improvement (CGI-I) is a 7-point rating of treatment response anchored by 1 ("very much improved) and 7 ("very much worse").

Blood will be collected including a sample for genetic testing. Then the first week of study drug and instructions on how to take it will be given. Please bring any unused study drug to on the next visit.

Visits 1/End of Week 1, 2/End of Week 2, 3/End of Week 4, 4/End of Week 8, 5/End of Week 12 Vital signs will be measured and a member of the research team will ask questions about current symptoms. Rating scales will be conducted assessing the symptoms.

Any unused study drug from the last visit will be collected and counted. The study doctor will ask about overall health and wellbeing. Please tell the study doctor about any problems encountered during the study. The next week's study drug will be given. Please bring any unused study drug to on the next visit.

Additional blood will be collected at visit 5.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder based on Structured Clinical Interview for DSM-IV (SCID)
* Hamilton Depression Rating Scale-24 (HRSD-24) score of 8-24.
* No antidepressant medication in past 3 months

Exclusion Criteria:

* Pregnancy/Breastfeeding/Reproductive age female not using contraception
* Schizophrenia or other psychotic disorders
* Bipolar Disorder
* Cluster B personality disorder
* Electroconvulsive Therapy (ECT) failure in past
* Concurrent ECT or repetitive transcranial magnetic stimulation (rTMS)
* Active substance abuse within past 6 months
* Use of antiepileptics
* Thyroid Stimulating Hormone (TSH) greater than 4
* Untreated Vitamin B12 deficiency (Vitamin B12 less than 400)
* Neurodegenerative disease or dementia (Mini Mental Status Examination (MMSE) less than or equal to 24)
* Suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale-24 | Week 12
  Clinician-administered questionnaire designed to assess the severity of depression in adults. It has been considered the gold standard for rating depression in clinical research.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Kanter, M.D., Principal Investigator — University of Florida
Locations (1):
- Shands Hospital Room HD-G-17, Gainesville, Florida, United States